CLINICAL TRIAL: NCT00006291
Title: A Phase II, Randomized, Partially Blinded Trial of Combinations of Potent Antiretroviral Therapy, HIV-Specific Immunizations, and Cycles of Interleukin-2 to Promote Efficient Control of Viral Replication
Brief Title: Safety and Effectiveness of Adding Either an HIV Vaccine, Interleukin-2, or Both to a Patient's Anti-HIV Drug Combination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: A5024; 10070 (Registry Identifier: DAIDS ES Registry Number); ACTG A5024; AACTG A5024
Record Dates: First submitted 2000-09-22; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Virus Replication; T-Lymphocytes; Lymphocyte Transformation; AIDS Vaccines; Anti-HIV Agents; Viral Load; Aldesleukin; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections | interventions — aldesleukin

INTERVENTIONS:
Biological: ALVAC(2)120(B,MN)GNP (vCP1452)
Drug: Aldesleukin

SUMMARY:
The purpose of this study is to see if adding an HIV vaccine (ALVAC-HIV vCP1452), IL-2 (interleukin-2, a protein found in the blood that helps boost the immune system), or both to anti-HIV-drug therapy is safe, tolerable, and effective in controlling viral load (level of HIV in the body). (This study has been changed to clarify drug name.) Anti-HIV drugs can help reduce a patient's viral load. However, HIV can still remain in CD4 cells (cells of the immune system that help fight infection). Combining an HIV vaccine, IL-2, or both with anti-HIV drugs may help reduce the number of HIV-infected cells.

DETAILED DESCRIPTION:
The most important goal for designing future therapeutic interventions is to understand the nature of persistent HIV infection in patients successfully treated with potent antiretroviral therapy and to develop strategies to promote the clearance of these reservoirs or at least long-term suppression of these reservoirs. If latently infected cells are able to persist for a long period (despite effective suppression of de novo infection) primarily because immune clearance is not being adequately stimulated by viral antigen, then HIV-specific immunization is a reasonable strategy to enhance the clearance of these cells. Stimulating effective HIV-specific cellular immune responses at a time when plasma viremia is maximally suppressed also may contribute to the long-term containment of HIV replication on potent antiretroviral therapy. A second component to be evaluated in this trial is whether broad, cyclical activation of T cells with IL-2 will increase the activation of HIV proviral gene expression and thereby render target cells susceptible to immune-mediated clearance. This pathogenesis-based clinical trial will explore the potential for these novel treatment strategies (HIV-specific immunization and IL-2, alone and in combination) to complement the effects of potent antiretroviral therapy by promoting more effective immunologic control of HIV-1 replication.

This study is divided into 3 steps.

STEP I: Patients continue to receive their stable potent antiretroviral therapy and are randomized to 1 of 4 arms:

Arm A: Vaccine placebo [AS PER AMENDMENT 08/23/01: ALVAC]; Arm B: Canarypox HIV-specific immunogen [AS PER AMENDMENT 08/23/01: ALVAC-HIV] (vCP1452); Arm C: 8-week cycles of IL-2 plus vaccine placebo [AS PER AMENDMENT 08/23/01: ALVAC]; Arm D: 8-week cycles of IL-2 plus canarypox HIV-specific immunogen [AS PER AMENDMENT 08/23/01: ALVAC-HIV] (vCP1452).

Patients receive vaccine (or vaccine placebo) injections at Weeks 0, 8, 16, 24, and 48. IL-2 injections are synchronized with vaccine injections. IL-2 is given open-label while vCP1452 is double-blinded. Patients must be on Step I for a minimum of 51 weeks [AS PER AMENDMENT 08/23/01: prior to entry into Step II].

STEP II: Patients stop study medications and interrupt potent antiretroviral therapy for [AS PER AMENDMENT 08/23/01: "6 to 16" has been replaced by the following text: a minimum of 12] weeks. Patients whose viral load during Step II remains [AS PER AMENDMENT 08/23/01: at or] below 5,000 copies/ml [AS PER AMENDMENT 08/23/01: and whose CD4 count is 200 cells/mm3 or more] are encouraged to remain off antiretroviral medications and continue viral-load monitoring for up to an additional 10 weeks. These patients are followed [AS PER AMENDMENT 08/23/01: "for up to 16 weeks" has been replaced by the following text: through Week 74] on Step II and must register to Step III only if their viral load increases to 50,000 copies/ml or greater, their CD4 count decreases to below 200 cells/mm3, or if their primary care physician recommends resuming antiretrovirals.

STEP III: Patients resume their original potent antiretroviral therapy regimen for 6 to 10 weeks and are monitored for a minimum of 6 weeks. If patients do not achieve a viral load below 50 copies/ml during those 6 weeks, they continue to be monitored for up to an additional 4 weeks until this degree of suppression is achieved with the same potent antiretroviral therapy regimen or another appropriate regimen.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible to enter this study if they:

* Are HIV-positive.
* Have taken the same anti-HIV drugs for at least 6 months prior to study entry. A change of 1 drug to another similar drug is allowed in certain cases.
* Have a viral load of less than 50 copies/ml at screening and pre-entry. The measurements must be within 45 days of study entry.
* Have a CD4 cell count of at least 350 cells/mm3 within 45 days prior to study entry.
* Agree to use effective methods of birth control during the study and for 12 weeks after.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Have or have had an AIDS-related illness (except Kaposi's sarcoma or Pneumocystis carinii pneumonia).
* Have had more than one potent antiretroviral regimen change due to virologic failure.
* Have a history of autoimmune disease with the exception of stable autoimmune thyroid disease.
* Have a history of allergy to eggs or other serious allergies.
* Have serious heart problems. Patients with high blood pressure controlled by blood pressure medication but no heart disease may be eligible for this study.
* Have cancer requiring chemotherapy.
* Have untreated thyroid disease. Patients who are on treatment and stable for at least 4 weeks before study entry are eligible.
* Have a serious central nervous system (CNS) disease or seizures, if these have been active within 1 year before study entry.
* Require certain heart medications for angina or arrhythmia.
* Are taking certain experimental anti-HIV drugs.
* Are taking certain drugs that may interfere with their anti-HIV-drug combination.
* Have taken drugs that might affect the immune system, within 4 weeks prior to study entry.
* Have taken IL-2 before.
* Have taken rifampin or rifabutin within 7 days before study entry if receiving indinavir.
* Have received therapy for an infection or any serious medical illness within 30 days before study entry.
* Have received immunizations within 30 days before study entry.
* Have received any HIV vaccine during the past year or at any time while on their present anti-HIV therapy.
* Work in close contact with canaries and are likely to have antibodies to the study vaccine prior to enrollment. (Patients with a pet canary may participate.)
* Abuse alcohol or drugs or have mental or learning problems.
* Are pregnant or breast-feeding.
* Have received abacavir or hydroxyurea within 8 weeks prior to study entry.
* Have a history of transplantation.
* (This study has been changed to reflect added criteria.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kilby, Study Chair; Ronald Mitsuyasu, Study Chair
Locations (26):
- United States (25):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Marin County Dept. of Health & Human Services, HIV/AIDS Program & Specialty Clinic, San Rafael, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - Univ. of Texas Medical Branch, ACTU, Galveston, Texas
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico